CLINICAL TRIAL: NCT02478814
Title: Evaluation of Protein Requirements in Active, Young Adult Males
Brief Title: Protein Requirements In Active Populations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Toronto (Other)
Collaborators: Ajinomoto Co., Inc. (Industry)
Responsible Party: Principal Investigator, Daniel Moore, Assistant Professor, University of Toronto
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: IAAO-YM
Record Dates: First submitted 2015-06-18; First posted 2015-06-23 (Estimated); Last update posted 2019-04-01 (Actual); Status verified 2019-03

CONDITIONS: Increased Metabolic Requirement; Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Active, Young Adult Males (Experimental): Subjects will receive different levels of amino acid intakes varying from 0.2 to 2.6 g/kg/day.
  Interventions: Dietary Supplement: Amino Acid Intake

INTERVENTIONS:
Dietary Supplement: Amino Acid Intake — Amino acid intakes will be varied at 0.2-2.6 g/kg/day

SUMMARY:
Protein requirements in active individuals have been suggested to be greater than the current recommended dietary allowance (RDA).

Nutritional requirements for dietary amino acids in adults have traditionally been determined utilizing the nitrogen balance technique, which is prone to underestimating protein requirements. As a result, there is a need to re-evaluate recommendations in order to characterize how dietary amino acid needs may be modulated by physical activity.

Recent studies using the minimally invasive indicator amino acid oxidation (IAAO) technique have suggested that protein requirements in young men are at least 50% higher than the RDA based on nitrogen balance data.

The purpose of this study is to measure the protein requirement in active, young adult males using the IAAO technique in the presence of a variable intensity exercise stimulus.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, active, young adult males who regularly participate in moderate-vigorous activity 5x per week, for a minimum of 1 hour
* A minimum score of 10 on the Beep Test (a measure of aerobic fitness)

Exclusion Criteria:

* Inability to meet health and physical activity guidelines according to the physical activity readiness questionnaire (PAR-Q+)
* Inability to adhere to any of the protocol guidelines (i.e. alcohol, caffeine consumption)
* Regular tobacco use
* Illicit drug use

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 7 (Actual)
Dates: Start 2015-04; Primary Completion 2016-06 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
13CO2 (carbon dioxide) excretion (μmol/kg/h) | 4 hours / study day

SECONDARY OUTCOMES:
13C-Phenylalanine Oxidation (μmol/kg/h) | 4 hours / study day

REFERENCES:
- [Derived] Packer JE, Wooding DJ, Kato H, Courtney-Martin G, Pencharz PB, Moore DR. Variable-Intensity Simulated Team-Sport Exercise Increases Daily Protein Requirements in Active Males. Front Nutr. 2017 Dec 21;4:64. doi: 10.3389/fnut.2017.00064. eCollection 2017. PMID 29312948